CLINICAL TRIAL: NCT01811641
Title: Epigenesis in Humans: Can Maternal Methyl-donor-deficient Diets Induce Epigenetic Alterations in Their Offspring?
Brief Title: Methyl-Donors and EpiGenetics in The Gambia
Acronym: MDEG
Status: Completed | Type: Observational
Sponsor: Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Matt Silver, MRC Senior Investigator Scientist, Medical Research Council
Other Study IDs: MRC-ING-MDEG
Record Dates: First submitted 2013-03-11; First posted 2013-03-14 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Aberrant DNA Methylation
Keywords: season of conception; maternal nutritional status; infant DNA methylation
MeSH Terms: interventions — Seasons; Eating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, buccal swab, hair follicles
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- maternal methyl-donors, infant epigenetics: women of reproductive age in rural Gambia, infants born to these women
  Interventions: Other: season, dietary intake

INTERVENTIONS:
Other: season, dietary intake

SUMMARY:
Accumulating evidence suggests that early-life nutrition can affect metabolism and thus increase the risk of disease in adulthood (e.g. type II diabetes and obesity). One possible mechanism to explain these effects is epigenetic variation at critical periods of development. Epigenetic variation describes non-inherited permanent alterations to an individuals DNA.

Recent work in mouse models has demonstrated that maternal nutritional status can affect such epigenetic processes such as DNA methylation and gene expression during embryonic development, with profound effects on outcomes. The investigators aim to study these processes in humans for the first time. The investigators will exploit the "experiment of nature" setting in The Gambia, i.e. fluctuation in diet according to season. During the 'hungry' season diets are known to be depleted in nutrients required for epigenetic gene regulation. Nutritional biomarkers in blood as well as the dietary intake will be measured in pregnant women according to season. A blood sample will also be taken from babies born to these women to determine whether there is a direct effect of diet on mothers' nutritional status and hence variation in DNA methylation patterns in their babies by season.

ELIGIBILITY:
Inclusion criteria women:

- women aged 18-45 years on 15th March 2009, resident in West Kiang

Exclusion criteria women:

* on contraception
* confirmed pregnancy at recruitment
* enrolment in any study other than the ENID (Early Nutrition and Immune Development) trial (ISRCTN49285450)
* suffering from severe anaemia (haemoglobin <7 g/dl) or known sickle cell disease

Inclusion criteria infants:

- born to the above women

Exclusion criteria infants:

- those known to be severely malnourished (weight-for-height Z-score < -3)

Ages: 1 Day to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: women of reproductive age in rural Gambia and their infants
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2009-01; Primary Completion 2012-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
DNA methylation of infants | infants: at 3-6 months of age
  Measurement of DNA methylation of infants recruited into the study, at 3-6 months of age.
  Measurement of blood biomarkers monthly after dietary assessment or in early pregnancy

SECONDARY OUTCOMES:
Blood biomarker status of women | monthly for 12 months or in early pregnancy
  Measurement of blood biomarkers monthly after dietary assessment or in early pregnancy

REFERENCES:
- [Result] Dominguez-Salas P, Moore SE, Baker MS, Bergen AW, Cox SE, Dyer RA, Fulford AJ, Guan Y, Laritsky E, Silver MJ, Swan GE, Zeisel SH, Innis SM, Waterland RA, Prentice AM, Hennig BJ. Maternal nutrition at conception modulates DNA methylation of human metastable epialleles. Nat Commun. 2014 Apr 29;5:3746. doi: 10.1038/ncomms4746. PMID 24781383
- [Result] Silver MJ, Kessler NJ, Hennig BJ, Dominguez-Salas P, Laritsky E, Baker MS, Coarfa C, Hernandez-Vargas H, Castelino JM, Routledge MN, Gong YY, Herceg Z, Lee YS, Lee K, Moore SE, Fulford AJ, Prentice AM, Waterland RA. Independent genomewide screens identify the tumor suppressor VTRNA2-1 as a human epiallele responsive to periconceptional environment. Genome Biol. 2015 Jun 11;16(1):118. doi: 10.1186/s13059-015-0660-y. PMID 26062908
- [Derived] Dominguez-Salas P, Moore SE, Cole D, da Costa KA, Cox SE, Dyer RA, Fulford AJ, Innis SM, Waterland RA, Zeisel SH, Prentice AM, Hennig BJ. DNA methylation potential: dietary intake and blood concentrations of one-carbon metabolites and cofactors in rural African women. Am J Clin Nutr. 2013 Jun;97(6):1217-27. doi: 10.3945/ajcn.112.048462. Epub 2013 Apr 10. PMID 23576045